CLINICAL TRIAL: NCT02579694
Title: Multicenter Retrospective-prospective Short-term Evaluation of the SLIC Screw System in Subjects Requiring Treatment for Acute Scapholunate Injury
Brief Title: Short Term Evaluation of SLIC Screw in Treatment of Scapholunate Injury
Status: Terminated | Type: Observational
Why Stopped: Difficulties finding subjects meeting enrollment criteria
Sponsor: Acumed, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 14013
Record Dates: First submitted 2015-10-15; First posted 2015-10-20 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Acute Scapholunate Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Acumed Scapholunate Intercarpal Screw — Evaluation of provisional fixation to allow biologic healing of the scapholunate interval
  Other Names: SLIC Screw

SUMMARY:
The purpose of this retrospective-prospective clinical evaluation is to determine whether the SLIC Screw System provides provisional fixation to allow biological healing of the scapholunate interval.

ELIGIBILITY:
Inclusion Criteria:

* Subjects willing and able to comprehend and sign Informed Consent
* Subjects who have received the SLIC screw as part of the treatment for scapholunate ligament repair or scapholunate reduction
* Subjects with acute scapholunate injury, classified with Garcia-Elias Stage 1-4, OR Geissler Stage 1-3
* Subjects >18 years of age at the time of surgery

Exclusion Criteria:

* Subject diagnosed with chronic scapholunate injury
* Subjects who underwent previous scapholunate procedure on the study wrist before implantation of the SLIC Screw System
* Subjects with active or latent infection at the time of surgery
* Subjects with sepsis at the time of surgery
* Subjects diagnosed with osteoporosis at the time of surgery
* Subjects with insufficient quantity and/or quality of bone
* Subjects with cartilage degeneration on the bones at the time of surgery
* Subjects with absence of potential for soft tissue healing at time of surgery, as documented by the investigator.
* Female Subjects known to be pregnant
* Subjects who were unable to follow postoperative care instructions, specifically, activity levels
* Subjects who are unable or unwilling to return for postoperative study visits

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients from selected sites with acute scapholunate injury fulfilling inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2015-09; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Comparison of reported VAS pain from preoperative to post-planned explantation | 12 months
  Planned removal of provisional device recommended between six and 9 months; 12-month analysis will capture time to planned removal.
Time to planned explantation is operationally defined as the time in days between device implantation and planned removal of an intact device | 12 months
The proportion of devices where removal is attributed to healing and not device failure | 12 months

SECONDARY OUTCOMES:
Radiographic evaluation of device integrity | 12 months
  Device integrity defined as no device breakage or separation
Radiographic evaluation of radiolucency | 12 months
Radiographic evaluation of osteolysis | 12 months
Complication rates over time | 12 months
Comparison of range of motion in degrees from preoperative values | 12 months
  Flexion, Extension, Radial Deviation, Ulnar Deviation
Comparison of grip strength in kg from preoperative values | 12 months
Comparison of reported VAS pain from preoperative values | 12 months
Subject satisfaction based on a five-point scale from preoperative | 12 months
Comparison of scapholunate angle from preoperative through radiographic evaluation | 12 months
Comparison of scapholunate joint space from preoperative through radiographic evaluation | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Unsell, MD, Principal Investigator — Community Hospital

REFERENCES:
- [Background] Zarkadas PC, Gropper PT, White NJ, Perey BH. A survey of the surgical management of acute and chronic scapholunate instability. J Hand Surg Am. 2004 Sep;29(5):848-57. doi: 10.1016/j.jhsa.2004.05.008. PMID 15465234
- [Background] Caloia M, Caloia H, Pereira E. Arthroscopic scapholunate joint reduction. Is an effective treatment for irreparable scapholunate ligament tears? Clin Orthop Relat Res. 2012 Apr;470(4):972-8. doi: 10.1007/s11999-011-1953-4. PMID 21732026
- [Background] Aviles AJ, Lee SK, Hausman MR. Arthroscopic reduction-association of the scapholunate. Arthroscopy. 2007 Jan;23(1):105.e1-5. doi: 10.1016/j.arthro.2006.07.013. Epub 2006 Oct 16. PMID 17210436
- [Background] Larson TB, Gaston RG, Chadderdon RC. The use of temporary screw augmentation for the treatment of scapholunate injuries. Tech Hand Up Extrem Surg. 2012 Sep;16(3):135-40. doi: 10.1097/BTH.0b013e318257595b. PMID 22913993
- [Background] Rosenwasser MP, Miyasajsa KC, Strauch RJ. The RASL procedure: reduction and association of the scaphoid and lunate using the Herbert screw. Tech Hand Up Extrem Surg. 1997 Dec;1(4):263-72. No abstract available. PMID 16609495
- [Background] Herbert TJ. Acute rotary dislocation of the scaphoid: a new technique of repair using Herbert screw fixation across the scapho-lunate joint. World J Surg. 1991 Jul-Aug;15(4):463-9. doi: 10.1007/BF01675642. PMID 1891931
- [Background] Opreanu RC, Baulch M, Katranji A. Reduction and maintenance of scapholunate dissociation using the TwinFix screw. Eplasty. 2009;9:e7. Epub 2009 Jan 29. PMID 19252680
- [Background] Cognet JM, Levadoux M, Martinache X. The use of screws in the treatment of scapholunate instability. J Hand Surg Eur Vol. 2011 Oct;36(8):690-3. doi: 10.1177/1753193411410154. Epub 2011 Jun 23. PMID 21700650
- [Background] Bhat AK, Kumar B, Acharya A. Radiographic imaging of the wrist. Indian J Plast Surg. 2011 May;44(2):186-96. doi: 10.4103/0970-0358.85339. PMID 22022028
- [Background] Loredo RA, Sorge DG, Garcia G. Radiographic evaluation of the wrist: a vanishing art. Semin Roentgenol. 2005 Jul;40(3):248-89. doi: 10.1053/j.ro.2005.01.014. No abstract available. PMID 16060116
- [Background] Garcia-Elias M. The treatment of wrist instability. J Bone Joint Surg Br. 1997 Jul;79(4):684-90. doi: 10.1302/0301-620x.79b4.14192. No abstract available. PMID 9250766